CLINICAL TRIAL: NCT05246969
Title: Detecting Sepsis in Patients With Severe Subarachnoideal Hemorrhage
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Principal Investigator, Goethe University
Other Study IDs: Sepsis in SAH
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Subarachnoid Hemorrhage; Subarachnoid Hemorrhage, Aneurysmal; Sepsis Syndrome; Sepsis; Sepsis, Severe; Sepsis Bacterial
Keywords: sequential organ failure assessment score
MeSH Terms: conditions — Subarachnoid Hemorrhage; Systemic Inflammatory Response Syndrome; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sepsis detection — The aim of the study was to observe whether the treating physicians were able to detect sepsis by strictly applying the recommended SOFA score.

SUMMARY:
The study aims to evaluate the suitability of the SOFA score implemented by the Sepsis 3 guideline to detect sepsis in patients suffering from subrarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

Critically ill patients suffering from moderate to severe subarachnoid hemorrhage (WFNS >2).

Exclusion Criteria:

children under the age of 18 years Patients with minor subarachnoid hemorrhage < WFNS stage 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe subarachnoid hemorrhage requiring intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Sepsis SOFA positive | up to 2 months
  Sepsis correctly detected by SOFA score (Sepsis-related organ failure assessment score, 0-24 points)
Sepsis SOFA negative | up to 2 months
  Sepsis not detected by SOFA score (Sepsis-related organ failure assessment score, 0-24 points)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Niederrad, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
The dataset will be published in an international journal. The data will be available upon reasonable request from the corresponding author